CLINICAL TRIAL: NCT03413059
Title: Thoracic Epidural Morphine Versus Triamcinolone Acetonide Analgesia in Flail Chest
Brief Title: Thoracic Epidural Analgesia in Flail Chest
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa hassanien hassanien bakr, assitent lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB1000
Record Dates: First submitted 2017-04-26; First posted 2018-01-29 (Actual); Last update posted 2018-01-29 (Actual); Status verified 2017-06

CONDITIONS: Flail Chest
MeSH Terms: conditions — Flail Chest | interventions — Morphine; Triamcinolone Acetonide; Triamcinolone

STUDY DESIGN:
Intervention Model Description: 1. Group (m): which will receive morphine dose 0.1mg /kg with 9 ml of 0.125 % bupivacaine with through epidural catheter in T 7-T10 .on admission. Then continuous epidural infusion of bupivacaine (0.1 mg.kg-1.h)
  2. Group (s) : will receive mixture consisting of 9 ml of 0.125 % bupivacaine with 80mg of triamcinolone ( 10 ml total volume) .through epidural catheter in-T7- T10 .on admission
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- morphine sulfate group (Active Comparator): patients in this arm will receive : morphine dose 0.1mg /kg with 9 ml of 0.25 % bupivacaine with through epidural catheter on admission Then continuous epidural infusion of bupivacaine (0.1 mg.kg-1.h) 1st 72 hours
  Interventions: Drug: Morphine Sulfate
- triamcinolone acetonide group (Active Comparator): patients in this arm will receive will receive a mixture of 9 ml of 0.125 % bupivacaine with 80mg of triamcinolone ( 10 ml total volume) through epidural catheter on admission
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: Morphine Sulfate — Thoracic Epidural morphine
  Other Names: morphine
  Arms: morphine sulfate group
Drug: Triamcinolone Acetonide — thoracic epidural triamcinolone acetonide
  Other Names: Triamcinolone
  Arms: triamcinolone acetonide group

SUMMARY:
The applicability of different thoracic epidural analgesia for patients with flail chest

DETAILED DESCRIPTION:
Pain due to traumatic rib fractures may be associated with increased morbidity and mortality. Fracture ribs cause severe pain that adversely affects patients' ability to cough and breathe deeply, that may lead to decreased ventilator efforts, atelectasis, pneumonia and finally respiratory failure. That further results in longer intensive care unit (ICU) and hospital length of stay and higher mortality. Effective pain relief, chest physiotherapy and respiratory care are the points of management. Effective analgesia enables the patient to breathe deeply, cough out the secretions and comply with chest physiotherapy. Multiple pain relief treatment options are available, such as oral analgesics, intravenous opioids, patient-controlled opioid analgesia, interpleural blocks, intercostals blocks, para vertebral blocks, and epidural analgesia Recent studies reported that epidural analgesia reduces morbidity after major thoracic, abdominal and vascular surgeries, but in patients with rib fractures, Successful treatment for rib fracture pain usually requires both pharmacologic and interventional approaches .Single modality treatment, which may incite respiratory depression, is suboptimal in these patients, many of whom already manifest a compromised respiratory system. Interventional procedures, while opioid sparing, carry their own inherent risks. Intercostals nerve blocks may not be feasible in the setting of multiple rib fractures, because of patient discomfort and the risk of local aesthetic toxicity. Use of an epidural catheter with continuous infusion of local anaesthetics and opioids may pose challenges in a community hospital setting, as 24 hours in-house coverage is often unavailable. While single-shot thoracic epidural steroid injections have been used for herniated intervertebral discs, herpes zoster pain, and post herpetic neuralgia (PHN), their use in patients with rib fracture pain has not been previously reported in the literature. An epidural steroid injection delivers steroids directly into the epidural space in the spine. Sometimes additional fluid (local aesthetic and/or a normal saline solution) is used to help 'flush out' inflammatory mediators from around the area that may be a source of pain ..Typically, a solution containing cortisone (steroid) with local aesthetic (lidocaine or bupivacaine), and/or saline is used.A steroid, or cortisone, is usually injected as an anti-inflammatory agent. Inflammation is a common component of many low back conditions and reducing inflammation helps reduce pain. Triamcinolone acetonide, Dexamethasone, and Methyl prednisolone acetate are commonly used steroids.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years.
* American Society of Anesthesiologists physical status 1 or 2.
* mentally competent and able to give consent for enrollment in the study

Exclusion Criteria:

* Patient refusal.
* Psychiatric disorder
* Patient younger than 18 years old
* Allergy to local anesthetics, systemic opioids (fentanyl, morphine)
* Impaired kidney functions and patient with coagulopathy will be also excluded.
* Chronic pain syndromes and patients with chronic opioid use defined as use of regular daily doses of systemic narcotics for the past 6 months prior to the surgery.
* BMI of 40 or more

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2018-07-01 (Estimated); Study Completion 2018-07-01 (Estimated)

PRIMARY OUTCOMES:
visual analogue score | 7 days
  mean visual analogue score (scale of 0 to 100) indicating the severity of pain

SECONDARY OUTCOMES:
ICU stay | 7 days
  from ICU admission to ICU discharge
chest infection | 7 days
  incidence of developing chest infection
hospital stay | 7 days
  length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Emad Z Saed, Principal Investigator — Lecturer. ansethsia department. Faculty of medicine .assuit unveristy.

IPD SHARING:
Plan to Share IPD: No